CLINICAL TRIAL: NCT06106594
Title: VOLT CE Mark Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10456
Record Dates: First submitted 2023-10-16; First posted 2023-10-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-03

CONDITIONS: Atrial Arrhythmia; Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Atrial Arrhythmia; Pulsed Field Ablation; Paroxysmal AF; PFA; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Main study enrollment will include up to 150 subjects, enrollment extension cohort will include up to 100 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Volt PFA Catheter Sensor Enabled (SE) (Experimental)
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — Pulsed field ablation using the Volt PFA System

SUMMARY:
This clinical investigation is intended to demonstrate safety and effectiveness of the Volt™ Pulsed Field Ablation (PFA) Catheter Sensor Enabled™, the Volt™ PFA Generator, Agilis™ NxT Steerable Introducer Dual-Reach™, and EnSite™ X EP System EnSite™ Pulsed Field Ablation Module (for simplicity of reference this device collection will hereafter be referred to as the Volt™ PFA system) for the treatment of symptomatic, recurrent, drug-refractory paroxysmal and persistent atrial fibrillation.

DETAILED DESCRIPTION:
The main study is a pre-market, prospective, single-arm, non-randomized, multicenter clinical study to demonstrate safety and effectiveness for the treatment of symptomatic, recurrent, drug-refractory Paroxysmal Atrial Fibrillation (PAF) and Persistent Atrial Fibrillation (PersAF). The main study design includes a feasibility sub-study in which additional imaging assessments will be collected in a small cohort of subjects to confirm acute safety of the Volt PFA System in humans.

The enrollment extension will include up to an additional 150 subjects enrolled with market-released or investigational devices, depending on enrollment geography.

ELIGIBILITY:
Inclusion Criteria:

1. Documented symptomatic PAF or PersAF. Documentation requirements are as follows:

   Paroxysmal:
   * Physician's note indicating recurrent self-terminating AF with ≥ 2 episodes of PAF within the 6 months prior to enrollment AND
   * One electrocardiographically documented PAF episodes within 12 months prior to enrollment.

   Persistent: Continuous AF sustained beyond 7 days and less than 1 year that is documented by
   * Physician's note, AND either
   * 24-hour Holter within 180-days prior to enrollment, showing continuous AF, OR
   * Two electrocardiograms (from any form of rhythm monitoring) showing continuous AF:

     * That are taken at least 7 days apart but less than 12 months apart
     * If electrograms are more than 12 months apart, there must be one or more Sinus Rhythm recordings in between or within 12 months prior to consent/enrollment
     * The most recent electrocardiogram must be within 180 days of enrollment.

   NOTE: Documented evidence of the AF episode must either be continuous AF on a 12-lead ECG or include at least 30 seconds of AF from another ECG device.
2. Plans to undergo a PVI catheter ablation procedure due to symptomatic PAF or PersAF and is refractory, intolerant, or contraindicated to at least one Class I-IV AAD medication
3. At least 18 years of age
4. Able and willing to comply with all trial requirements including pre-procedure, post- procedure, and follow-up testing and requirements
5. Informed of the nature of the trial, agreed to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical trial site.

Exclusion Criteria:

1. Previously diagnosed long-standing persistent atrial fibrillation (AF greater than 1 year in duration)
2. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, electrolyte imbalance, severe untreated sleep apnea, and other major surgical procedures in the preceding 90 days
3. Participant known to require ablation beyond PVI at the time of consent (Main study only)
4. Known presence of cardiac thrombus
5. Left atrial diameter ≥ 5.5 cm (anteroposterior diameter)
6. Left ventricular ejection fraction < 35% as assessed with echocardiography within 180 days of index procedure
7. New York Heart Association (NYHA) class III or IV heart failure
8. Body mass index > 40 kg/m2
9. Pregnant, nursing, or planning to become pregnant during the clinical investigation follow-up period
10. Patients who have had a ventriculotomy or atriotomy within the preceding 28 days of procedure,
11. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 90 days
12. Unstable angina
13. Stroke or TIA (transient ischemic attack) within the last 90 days
14. Heart disease in which corrective surgery is anticipated within 180 days after procedure
15. History of blood clotting or bleeding abnormalities including thrombocytosis, thrombocytopenia, bleeding diathesis, or suspected anti-coagulant sate
16. Contraindication to long term anti-thromboembolic therapy
17. Patient unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
18. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
19. Previous left atrial surgical or catheter ablation procedure (including LAA closure device)
20. Presence of any condition that precludes appropriate vascular access
21. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).
22. Previous tricuspid or mitral valve replacement or repair
23. Patients with prosthetic valves
24. Patients with a myxoma
25. Patients with an interatrial baffle or patch as the transseptal puncture could persist and produce an iatrogenic atrial shunt
26. Stent, constriction, or stenosis in a pulmonary vein
27. Rheumatic heart disease
28. Hypertrophic cardiomyopathy
29. Diagnosed with amyloidosis or atrial amyloidosis
30. Active systemic infection
31. Renal failure requiring dialysis
32. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
33. Presence of an implantable therapeutic cardiac device including permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) or planned implant of such a device for any time during the follow-up period. Presence of an implantable loop recorder is acceptable as long as it is removed prior to insertion of the investigational device.
34. Presence of an implanted LAA closure device or plans to have an LAA closure device implanted during the follow-up period
35. Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this clinical trial without pre-approval from this study Sponsor
36. Unlikely to survive the protocol follow up period of 12 months
37. Presence of other medical, anatomic, comorbid, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
38. Individuals without legal authority
39. Individuals unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of subjects experiencing a device and/or procedure-related serious adverse event with onset within 7-days of any ablation procedure that uses the Volt PFA System. | 7-days
  Serious adverse events are defined as:
  * Atrio-esophageal fistula
  * Cardiac tamponade/perforation
  * Death
  * Heart block
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve injury resulting in permanent diaphragmatic paralysis
  * Pulmonary edema
  * Pulmonary vein stenosis
  * Stroke/cerebrovascular accident
  * Thromboembolism
  * Transient ischemic attack
  * Vagal nerve injury/gastroparesis
  * Major vascular access complications / major bleeding events
  * Device and/or procedure related cardiovascular and/or pulmonary adverse event that prolongs hospitalization for more than 48 hours (excluding hospitalization solely for arrhythmia recurrence or non-urgent cardioversion)
Acute procedural effectiveness summarized as the rate of pulmonary veins treated with the Volt PFA system that are isolated at the end of the index ablation procedure. | During procedure
  Acute procedural failure for each pulmonary vein is defined as any of the following:
  1. Inability to isolate a pulmonary vein at the end of the index ablation procedure. Isolation will be assessed via confirmation of electrical isolation in each ablated pulmonary vein after a minimum waiting period of 20 minutes via entrance block at a minimum. Touch-up ablation to achieve isolation will be allowed for any pulmonary vein reconnection detected during the index procedure with the investigational catheter (to the maximum delivery allowed per vein) and will not be considered a failure.
  2. Any use of a non-study ablation device for pulmonary vein isolation.
Long-term 6-month effectiveness summarized as the rate of freedom from documented AF/AFL/AT episodes of >30 seconds duration after the index ablation procedure through 6 months of follow-up. | 6 months
  The situations in which subjects will be considered long-term effectiveness endpoint failures:
  * Acute procedural failure
  * Any use of a non-study ablation device for pulmonary vein isolation or to deliver ablation lesions in the left atrium during the index procedure or during the first repeat procedure.
  * If documented AF/AFL/AT recurrence occurs at any time after the blanking period
  * If subject requires a repeat procedure for the treatment of AF, non-CTI-dependent AFL, or AT after the blanking period or a second repeat AF ablation procedure at any time after the index ablation procedure.
  * Any use of a new class I or III AAD for AF after the blanking period.
  * Any use of a class I or III AAD for AF at a dose higher than the historical maximum dose for the subject after the blanking period.
  * If the subject requires a cardioversion for the treatment of AF/AFL/AT after the blanking period
  * Surgical treatment of AF/AFL/AT post index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, Study Director — Abbott
Locations (16):
- Australia (4):
  - The Prince Hospital, Chermside, Queensl
  - Royal Adelaide Hospital, Adelaide, Saustrl
  - Monash Health, Clayton, Victoria
  - Royal Melbourne Hospital - City Campus, Parkville, Victoria
- A. ö. Krankenhaus der Elisabethinen Linz, Linz, UPR AUS, Austria
- Belgium (2):
  - UZ Brussel, Brussels, Brussels Capital
  - AZ Sint Jan, Bruges, Wflndrs
- Nemocnice Na Homolce, Prague, Cbohmia, Czechia
- Germany (3):
  - Medizinische Einrichtungen der Universität zu Köln, Cologne, N. RHIN
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck, Schlesw
  - Universitätsmedizin Berlin - Charité Campus Mitte (CCM), Berlin, State of Berlin
- Az. Osp.Universitaria Osp.Riuniti Umberto I-Lancisi-Salesi, Ancona, The Marches, Italy
- UMC Utrecht, Utrecht, Utrecht, Netherlands
- Hospital Universitari i Politècnic La Fe, Valencia, Valencia, Spain
- Hôpital Cantonal Universitaire de Geneva, Geneva, Canton of Geneva, Switzerland
- St. Bartholomew's Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tilz RR, Chierchia GB, Gunawardene M, Sanders P, Haqqani H, Kalman J, Healy S, Purerfellner H, Neuzil P, Asensi JO, Loh P, Reddy VY, Knecht S, Jesser E, Dirckx N, Miller A, Walker D, Lakkireddy D. Safety and effectiveness of the first balloon-in-basket pulsed field ablation system for the treatment of atrial fibrillation: VOLT CE Mark Study 6-month results. Europace. 2025 Mar 28;27(4):euaf072. doi: 10.1093/europace/euaf072. PMID 40163671
- [Result] Sanders P, Healy S, Emami M, Kotschet E, Miller A, Kalman JM. Initial clinical experience with the balloon-in-basket pulsed field ablation system: acute results of the VOLT CE mark feasibility study. Europace. 2024 May 2;26(5):euae118. doi: 10.1093/europace/euae118. PMID 38701222